CLINICAL TRIAL: NCT07014631
Title: A Phase II Dose-Finding Study to Evaluate the Efficacy and Safety of Oral SSS17 Capsules for Anemia in Non-Dialysis Chronic Kidney Disease Patients
Brief Title: Phase II Dose-Finding of Oral SSS17 for Anemia in Non-Dialysis CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSS-SSS17-RA-II-01
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Anemia in Pre-Dialysis Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSS17 (Experimental): The SSS17 treatment arm comprises three dose levels: the first two dose levels will have an 8-week treatment duration, while the third dose level will extend to 24 weeks. At each dose level, participants will be allocated in a 4:1 ratio (SSS17:placebo) for enrollment
  Interventions: Drug: SSS17
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSS17 — The SSS17 treatment arm comprises three dose levels: the first two dose levels will have an 8-week treatment duration, while the third dose level will extend to 24 weeks. At each dose level, participants will be allocated in a 4:1 ratio (SSS17:placebo) for enrollment.
  Arms: SSS17
Drug: Placebo — At each dose level, participants will be allocated in a 4:1 ratio (SSS17:placebo) for enrollment.Placebo recipients will undergo weekly dosing identical to the active treatment group within their assigned dose cohort.
  Arms: placebo

SUMMARY:
This study primarily evaluates the efficacy and safety of oral SSS17 capsules in treating anemia in patients with non-dialysis chronic kidney disease, as well as the pharmacokinetic and pharmacodynamic (PK/PD) characteristics of different doses of SSS17 capsules for anemia treatment in this patient population.

DETAILED DESCRIPTION:
This dose-finding study comprises three distinct dosing cohorts:cohort 1-3 once weekly . Each cohort will enroll patients at a 4:1 ratio (SSS17:placebo), allocating 32 subjects to active treatment and 8 to placebo control per group. The total planned enrollment is 120 non-dialysis chronic kidney disease (CKD) patients with anemia.

The trial will initiate with Cohort 1. Dosing regimens for subsequent cohorts may be modified based on predefined pharmacokinetic (PK), pharmacodynamic (PD), and safety evaluations from preceding cohorts, including potential adjustments to dose levels and/or administration frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Non-dialysis CKD patients aged 18-75 years.
2. Screening eGFR <60 mL/min/1.73 m² .
3. Mean Hb ≥7.0 g/dL and <10.0 g/dL .
4. Agreement to use medically acceptable contraception from ICF signing until 6 months post-trial.

Exclusion Criteria:

1. Hypoxia-inducible factor prolyl hydroxylase inhibitors within 5 weeks pre-randomization.
2. Erythropoiesis-stimulating agents, androgens, IV iron , or other anemia drugs within 6 weeks pre-randomization.
3. Blood donation/transfusion within 3 months
4. Transferrin saturation ≤20% and ferritin ≤100 μg/L at screening.
5. Uncorrected folate or vitamin B12 deficiency pre-randomization.
6. Systolic BP >170 mmHg, diastolic BP >110 mmHg.
7. iPTH >500 pg/mL.
8. Acute/chronic pancreatitis or amylase/lipase >3×ULN.
9. NYHA Class III/IV heart failure or significant arrhythmias .
10. Proliferative diabetic retinopathy, macular edema, or other neovascular retinal disorders requiring treatment.
11. Active HBV, HCV, HIV, or clinically significant uncontrolled infections.
12. Current/pplanned dialysis, prior nephrectomy, polycystic kidney disease, or hemochromatosis.
13. Organ transplant recipient/candidate，Participation in other drug trials within 3 months，Substance abuse history.
14. Pregnancy, lactation, or refusal of contraception.
15. Hypersensitivity to study drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 86 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin from baseline | Week7~Week9

SECONDARY OUTCOMES:
Weekly changes in hemoglobin from baseline | Week2~Week9
Proportion of subjects achieving hemoglobin response (≥10 g/dL) | Week7~Week9
Cumulative proportion of subjects achieving both Hb increase ≥10 g/L and Hb level ≥100 g/L | Week9

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided